CLINICAL TRIAL: NCT03970356
Title: The Improving Rational Prescribing for Urinary Tract Infections in Frail Elderly (ImpresU) Project - Work Package 2 (WP2): a Cluster Randomised Multifaceted Antibiotic Stewardship Intervention Study
Brief Title: Improving Antibiotic Prescribing for Urinary Tract Infections in Frail Elderly
Acronym: ImpresU-WP2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cees Hertogh (Other)
Collaborators: UMC Utrecht (Other); Medical University of Lodz (Other); University of Oslo (Other); Vastra Gotaland Region (Other Government); Göteborg University (Other)
Responsible Party: Sponsor-Investigator, Cees Hertogh, Prof. dr., Amsterdam UMC, location VUmc
Organization: Amsterdam UMC, location VUmc (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2005035; 25 (2017) (Other Grant/Funding Number: JPIAMR); 549003002 (Other Grant/Funding Number: ZonMW, Netherlands); 2017/25/Z/NZ7/03024 (Other Grant/Funding Number: National Science Centre, Poland); 2017-05975 (Other Grant/Funding Number: The Swedish Research Council); 284253 (Other Grant/Funding Number: The Research Council of Norway)
Record Dates: First submitted 2019-05-26; First posted 2019-05-31 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Urinary Tract Infections
Keywords: cluster randomized trial; antibiotic stewardship; frail elderly
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Intervention Model Description: The investigators will perform a pragmatic cluster randomised controlled trial (cRCT). The targeted population consists of frail elderly residents of residential care homes and nursing homes attended by general practitioners. The clusters (care home + general practitioners) are assigned to intervention- or control group. In the intervention group, an antibiotic stewardship intervention is actively implemented at the level of the general practitioners and caregivers in the homes.
  The study has two measurement periods; a baseline period (5 months) and a follow-up period (7 months). In between there is an implementation period in which the intervention (i.e. active implementation) is started in the intervention homes [no measurements are taken].
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention (Experimental): The antibiotic stewardship intervention will encourage to prescribe according to the latest relevant UTI guidelines which promote more restrictive use of antibiotics in case of non-specific symptoms.
  Interventions: Other: antibiotic stewardship intervention
- control (No Intervention): Usual care

INTERVENTIONS:
Other: antibiotic stewardship intervention — The intervention is multifaceted, consisting of the implementation of an algorithm for restrictive use of antibiotics as proposed in recent guidelines (Verenso, Dutch guideline), tailored in close collaboration with local stakeholders to the specific implementation setting, by means of a modified participatory-action research (PAR) approach. To support the process of intervention-tailoring and -implementation, a toolbox comprising of materials, aids and actions is developed to be used at the discretion of the local stakeholders to support implementation of the algorithm.The algorithm is congruent with the Swedish and Norwegian guidelines, which also promote more restrictive use of antibiotics in case of non-specific symptoms, even though the algorithm is more detailed.
  Arms: intervention

SUMMARY:
The purpose of this study is to determine whether a tailored multifaceted antibiotic stewardship intervention reduces antibiotic use for urinary tract infections in residential care homes and nursing homes attended by general practitioners. This will be evaluated in a pragmatic cluster randomised controlled trial using a modified community-based participatory action research approach.

DETAILED DESCRIPTION:
Rationale:

Almost 60% of antibiotics in frail elderly is prescribed for alleged UTI. About half of the antibiotics for UTI in this population are prescribed for non-specific signs and symptoms; a substantial part of these prescriptions might not be necessary.

Research question:

Does a tailored multifaceted antibiotic stewardship intervention reduce antibiotic use for UTI in residential care homes and nursing homes attended by general practitioners (GPs)?

Study design, setting and population:

A pragmatic cluster randomised controlled trial using a modified community-based participatory action research approach. In the intervention group the latest UTI guidelines (which are standard care) are actively implemented at the level of the GP/caregivers. Residents ≥ 70 year with ADL dependency from 34 care homes + attending GP practices will participate in Norway, Sweden, Poland and the Netherlands.

Methods:

The study has two measurement periods; a baseline period (5 months) and a follow-up period (7 months). In between the antibiotic stewardship intervention will be tailored and implemented in intervention practices. GPs will prospectively register suspected UTIs on standardized registration forms and (study) nurses/assistants will follow-up patients at day 7 and day 21 for each UTI.

Patients will be enrolled prior to the start of the study.

* June-August 2019: patient are recruited, informed consent is obtained, baseline characteristics of patients are recorded
* Sept 2019: study starts (from this moment onwards, the outcomes are being assessed).

Data analysis:

The primary analysis will be to assess the number of prescriptions of antibiotics for suspected UTI in the follow-up period, correcting for the baseline period and controlled for pre-specified confounders, using a generalized linear mixed model for Poisson distributions.

ELIGIBILITY:
Inclusion Criteria:

* physical and/or mental disabilities and ADL dependency requiring residential care or nursing home care
* attended by general practitioners
* not on continuous prophylactic antibiotic use

Exclusion Criteria:

* in hospice-care
* very limited life expectancy (≤1 month)
* no longer wish to participate
* start continuous antibiotic (prophylaxis)
* die or move away from the residential care home / nursing home

If patients are excluded within 2 months after inclusion, they will be taken out of the study. In other words: patients need to be included for at least 2 months to contribute data to the study.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1146 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-07-21 (Actual); Study Completion 2021-07-21 (Actual)

PRIMARY OUTCOMES:
UTI prescriptions | Assessed during the 7-month follow-up period
  Number of prescriptions of antibiotics for suspected urinary tract infections expressed per patient-year

SECONDARY OUTCOMES:
Incorrect UTI prescriptions | Assessed during the 7-month follow-up period
  Number of incorrect prescriptions of antibiotics for suspected UTI expressed per patient-year
UTI suspicions | Assessed during the 7-month follow-up period
  Incidence of suspected UTI expressed per patient-year
Complications | Assessed during the 7-month follow-up period
  Incidence of complications: delirium, pyelonephritis, sepsis and renal failure within 21 days after each UTI suspicion
Hospital referral | Assessed during the 7-month follow-up period
  Incidence of referral to a hospital within 21 days after each UTI suspicion
Hospital admission | Assessed during the 7-month follow-up period
  Incidence of hospital admission within 21 days after each UTI suspicion
Mortality | Assessed during the 7-month follow-up period
  Mortality
Mortality after UTI suspicion | Assessed during the 7-month follow-up period
  Mortality within 21 days after each UTI suspicion
UTI prescriptions in office hours | Assessed during the 7-month follow-up period
  Number of prescriptions of antibiotics for suspected UTI in office hours expressed per patient-year

CONTACTS AND LOCATIONS:
Overall Officials: Cees MP Hertogh, prof. dr., Principal Investigator — Amsterdam UMC, location VUmc; Theo JM Verheij, prof. dr., Principal Investigator — UMC Utrecht; Maciek Godycki-Cwirko, prof.dr., Principal Investigator — Medical University of Lodz; Morten Lindbæk, prof. dr., Principal Investigator — University of Oslo; Pär-Daniel Sundvall, MD PhD, Principal Investigator — Göteborg University
Locations (4):
- University Medical Center Utrecht, Utrecht, Netherlands
- University of Oslo, Oslo, Norway
- Medical University of Lodz, Lodz, Poland
- Research and Development Primary Health Care, Region Västra Götaland, Borås, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hartman EAR, Groen WG, Heltveit-Olsen SR, Lindbaek M, Hoye S, Lithen SS, Sundvall PD, Sundvall S, Snaebjornsson Arnljots E, Gunnarsson R, Kowalczyk A, Godycki-Cwirko M, van de Pol AC, Platteel TN, Monnier AA, Verheij TJM, Hertogh CMPM. Implementation of a tailored multifaceted antibiotic stewardship intervention to improve antibiotic prescribing for urinary tract infections in frail older adults (ImpresU) in four European countries: a process evaluation alongside a pragmatic cluster randomized controlled trial. Trials. 2024 Oct 18;25(1):691. doi: 10.1186/s13063-024-08545-4. PMID 39425170
- [Derived] Hartman EAR, van de Pol AC, Heltveit-Olsen SR, Lindbaek M, Hoye S, Lithen SS, Sundvall PD, Sundvall S, Arnljots ES, Gunnarsson R, Kowalczyk A, Godycki-Cwirko M, Platteel TN, Groen WG, Monnier AA, Zuithoff NP, Verheij TJM, Hertogh CMPM. Effect of a multifaceted antibiotic stewardship intervention to improve antibiotic prescribing for suspected urinary tract infections in frail older adults (ImpresU): pragmatic cluster randomised controlled trial in four European countries. BMJ. 2023 Feb 22;380:e072319. doi: 10.1136/bmj-2022-072319. PMID 36813284
- [Derived] Hartman EAR, Groen WG, Heltveit-Olsen SR, Lindbaek M, Hoye S, Sundvall PD, Gunnarsson R, Skoglund I, Snaebjornsson Arnljots E, Godycki-Cwirko M, Kowalczyk A, Platteel TN, Zuithoff NPA, Monnier AA, Verheij TJM, Hertogh CMPM, van de Pol AC. Multifaceted antibiotic stewardship intervention using a participatory-action-research approach to improve antibiotic prescribing for urinary tract infections in frail elderly (ImpresU): study protocol for a European qualitative study followed by a pragmatic cluster randomised controlled trial. BMJ Open. 2021 Oct 7;11(10):e052552. doi: 10.1136/bmjopen-2021-052552. PMID 34620666